CLINICAL TRIAL: NCT02853812
Title: Tinnitus Related Cerebral Activities: Personalised Approach of the Tinnitus Treatment
Brief Title: Tinnitus Related Cerebral Activities
Acronym: ACCELA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of inclusion period
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8847
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Tinnitus
Keywords: tinnitus; residual inhibition
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single sided tinnitus (Other): patients with single sided tinnitus on which functional brain MRI is assessed
  Interventions: Other: Functional brain MRI

INTERVENTIONS:
Other: Functional brain MRI — Sound evoked functional MRI assessment on patients with single sided tinnitus

SUMMARY:
The proposed research is to identify the brain areas activated or deactivated by tinnitus in humans. The identification of these areas is expected to be able to treat tinnitus refractory to traditional therapies by methods of brain stimulation. Furthermore, this technique would be very useful to verify the effectiveness of any treatment to relieve tinnitus.

The brain activation measured during fMRI will be performed in a position of rest, after inhibition of tinnitus, and after application of a sound that does not inhibit tinnitus. This comparison will identify specific brain areas activated or deactivated by tinnitus.

DETAILED DESCRIPTION:
1. What is the purpose of the research?

   The proposed research is to identify the brain areas activated or deactivated by tinnitus in humans.

   The identification of these areas is expected to be able to treat tinnitus refractory to traditional therapies by methods of brain stimulation.

   Furthermore, this technique would be very useful to verify the effectiveness of any treatment to relieve tinnitus.
2. What is the methodology?

   This is a diagnosis based on functional brain imaging with MRI (fMRI).

   The study will be conducted in 30 subjects with unilateral tinnitus, stable lesion of origin and can be inhibited by masking sound.

   The brain activation measured during fMRI will be performed in a position of rest, after inhibition of tinnitus, and after application of a sound that does not inhibit tinnitus.

   This comparison will identify specific brain areas activated or deactivated by tinnitus.
3. What are the expected benefits?

Direct individual benefit could possibly be met by participants in this study. Indeed, the determination of a masking noise can afford to set up a masking system to reduce the tinnitus if the patient wishes.

Moreover, in case of identification of brain areas activated or inactivated by tinnitus in a subject, it may propose to carry out a transcranial magnetic brain stimulation of the area in an attempt to relieve the tinnitus, according to the stimulation protocols to date for tinnitus.

This will achieved a personalized approach to treating tinnitus.

Besides the expected individual benefit, other expected benefits are collective order, given the highly variable success rates, but generally limited treatments against tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Age limits to > 18 years and < 70 years
* Voluntary study participation
* Unhurt of any acute or chronic pathology of the ear (except tinnitus and a possible deafness of perception in the limits fixed below) on the basis of the interrogation and of the clinical examination
* presenting a single sided tinnitus
* Presenting on the side of the tinnitus a phenomenon of residual inhibition with a duration of total disappearance of the tinnitus of more than 30 seconds
* easily reached
* informed consent signed
* Affiliation or recipient with the mode of social security

Exclusion Criteria:

* Subjects incapable to understand the nature and the purposes of the study and/or having difficulty of communication with the investigator
* majors protected by the law or privated of liberty by judiciary or administrative decision
* pregnant woman
* instable tinnitus (difference upper than 3 on mean of the EVA realised during the 5 days before the inclusion)
* insufficient tinnitus intensity (mean of the EVA realised during the 5 days before the inclusion<4)
* Anomaly of the external or average ear
* Tinnitus attributed to a clearly identified retro-cochlear origin
* Deafness of transmission of more than 15 dB on the tonal audiometry
* Deafness of perception of more than 60 dB in average hearing loss (arithmetic mean) on the frequencies of 0,5-1-2 and 4 kHz.
* Renowned ototoxic treatment during the duration of the protocol (malaria medicines, ototoxic chemotherapy, ototoxic antibiotic treatment),
* Pursuit of a noise exposure of strong intensity with title professional and/or of leisure, dental treatment with use of engine or turbine, during the duration of the protocol.
* Contraindication in the examination MRI (pacemaker, port of surgical clips in the cervico-cephalic region or implanted medical surgical material susceptible to mobilize under the influence of magnetic gradients, foreign body intraocular, pieces of shrapnel at the cervico-cephalic level (possibility of artefact), claustrophobia, pregnancy of less than 3 months)
* History of cranial trauma with encephalic infringement(achievement), ischemic cerebrovascular accident or intracerebral bruise.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02-05 (Actual); Primary Completion 2015-08-27 (Actual); Study Completion 2015-08-27 (Actual)

PRIMARY OUTCOMES:
Measure of the BOLD activity by MRI | 6 months
  Measure is done by MRI

SECONDARY OUTCOMES:
Measure of the BOLD activity on resting state by MRI | 6 months
  Measure is done by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Venail, MD PhD, Study Chair — CHU de Montpellier

IPD SHARING:
Plan to Share IPD: No